CLINICAL TRIAL: NCT04614350
Title: A Pilot Study For Healing And Safety Outcomes In Creating Site Appropriate Keratinized Tissue Comparing Markman Biologics Microsurfaced ADM And AlloDerm ADM
Brief Title: Pilot Study for Healing and Safety Outcomes in Gingival Recession
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: CellTherX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB2020-01
Record Dates: First submitted 2020-09-02; First posted 2020-11-04 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, within subjects-controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-Active (Experimental): Markman Biologics microsurfaced ADM
  Interventions: Biological: Markman Biologics Microsurfaced ADM
- B-Control (Active Comparator): AlloDerm ADM
  Interventions: Biological: AlloDerm

INTERVENTIONS:
Biological: Markman Biologics Microsurfaced ADM — an ADM which has been scored (microsurfaced)
  Arms: A-Active
Biological: AlloDerm — AlloDerm tissue matrix
  Arms: B-Control

SUMMARY:
Prospective, randomized, within subjects-controlled design

DETAILED DESCRIPTION:
The objective of this trial is to evaluate clinical healing outcomes of microsurfaced cadaveric ADM (Markman Biologics) used in sites with < 1 mm of attached gingiva requiring soft tissue grafting without root coverage as compared to control cadaveric ADM (AlloDerm, LifeCell) over 180-day post-op period. During the treatment period, each site will be monitored for soft tissue healing and augmentation of keratinized tissue width. All subjects will be seen at post-op day 7, 14, 30, 90, and 180.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or Legally Authorized Representative (LAR)
2. Patients with ≥2 non-adjacent teeth in the same jaw presenting with ≤ 1mm attached gingiva that requires soft tissue grafting without the need for root coverage
3. Patients with good oral hygiene as indicated by presence of minimal plaque and absence of material alba and calculus.
4. ≥ 18 and ≤ 75 years of age
5. Sexually active subjects (both men and women) who agree to use acceptable contraceptive methods for the duration of the study.

Exclusion Criteria:

1. Vestibule depth <7mm from the base of recession
2. Systemic condition, such as uncontrolled diabetes mellitus, HIV, cancer, or bone metabolic disease that could compromise wound healing
3. Treatment with systemic corticosteroids, immunosuppressive agents, radiation therapy, or chemotherapy within 2 months of enrollment in the study
4. Acute infection lesions in intended grafting sites
5. Received intravenous or intramuscular bisphosphonates
6. Tobacco use within 3 months of enrollment or for the duration of the study
7. Only molar teeth suitable for soft tissue grafting (molars may be treated but not assigned as the study tooth)
8. Miller grade ≥2 mobility on grafting sites or adjacent teeth
9. Known hypersensitivity to bovine collagen or iodine (shellfish allergy)
10. Previous treatment with an advanced biologic at sites selected fro grafting or the adjacent teeth
11. Pregnant or nursing female subjects; women of child-bearing potential must have a negative urine pregnancy test.
12. Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
13. Active alcohol or substance abuse (including marijuana, THC, CBD oils and products) in the opinion of the investigator that could impair the subject's participation in the study.
14. Any medical condition or co-morbidity that in the opinion of the investigator, would prevent successful participation in the study
15. Known allergies to Cefoxitin, Gentamycin, Lincomycin, Polymyxin B, Vancomycin, or any antibiotic in these same classes.
16. Known allergy to Polysorbate 20

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To compare graft healing at post-op day 14 between Markman Biologics Microsurfaced ADM (Active) and AlloDerm ADM (Control) as assessed by color | Day 14 post op
  tissue color
To compare graft healing at post-op day 14 between Markman Biologics Microsurfaced ADM (Active) and AlloDerm ADM (Control) as assessed by texture | Day 14 post op
  graft texture assessed as smooth, stippled, rolled, or other and as more firm, equally firm, less firm
To compare graft healing at post-op day 14 between Markman Biologics Microsurfaced ADM (Active) and AlloDerm ADM (Control) as assessed by inflammation | Day 14 post op
  tissue inflammation using a score of 0 (normal) to 4 (severe)
To compare graft healing at post-op day 14 between Markman Biologics Microsurfaced ADM (Active) and AlloDerm ADM (Control) as assessed by graft failure | Day 14 post op
  graft failure by no evidence of keratinized tissue width
To compare graft healing at post-op day 14 between Markman Biologics Microsurfaced ADM (Active) and AlloDerm ADM (Control) as assessed by graft loss | Day 14 post op
  graft loss

SECONDARY OUTCOMES:
Graft Healing | 180 days
  graft healing is assessed by by multiple means
Clinical Attachment level | 180 days
  change in measured clinical attachment level from baseline to Day 180
Change in Probing depths | 180 days
  change in measurement of probing depth from baseline to Day 180
Change in recession | 180 days
  change in measurement of recession from baseline to Day 180
Change in keratinized tissue | 180 days
  change in measurement of keratinized from baseline to Day 180
Change in gingival attachment | 180 days
  change in measurement of gingival attachment from baseline to Day 180
Healing as assessed by histological analysis | 90 days post op
  analysis by H&E staining of biopsied tissue
Assessment of Infection through 180 days | 180 days
  infection assesse by redness, swelling, pus, fevers, chills
Occurrence of AEs/SAEs | through 180 days
  Adverse events/Serious adverse events reported by site
Subject Discomfort | through 180 days
  Subject discomfort will be assessed using a single questionnaire containing questions on pain and the need for anti-inflammatory and/or pain meds.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Heard, DDS, Study Director — The McGuire Institute
Locations (1):
- Perio Health Professionals, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a single site study so data will not be other PIs to share the data with.